CLINICAL TRIAL: NCT02547077
Title: Use of 2-octylcyanoacrylate (Dermabond) Versus 5-0 Fast Absorbing Gut During Cutaneous Wound Closure: a Randomized Evaluator Blinded Split Wound Comparative Effectiveness Trial
Brief Title: Use of 2-octylcyanoacrylate (Dermabond) Versus 5-0 Fast Absorbing Gut During Cutaneous Wound Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 774875
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Wound Closure Techniques
MeSH Terms: interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wound Closure with 2-octylcyanoacrylate (Experimental): One side of the patient's wound defect will be assigned to wound closure with 2-octylcyanoacrylate liquid bonding agent).
  Interventions: Procedure: Wound Closure with 2-octylcyanoacrylate; Procedure: Wound Closure with 5-0 Fast Absorbing Gut Sutures
- Wound Closure with 5-0 Fast Absorbing Gut (Active Comparator): One side of the patient's wound defect will be assigned to wound closure with 5-0 fast absorbing gut sutures.
  Interventions: Procedure: Wound Closure with 2-octylcyanoacrylate; Procedure: Wound Closure with 5-0 Fast Absorbing Gut Sutures

INTERVENTIONS:
Procedure: Wound Closure with 2-octylcyanoacrylate
Procedure: Wound Closure with 5-0 Fast Absorbing Gut Sutures

SUMMARY:
The purpose of this study is to determine whether the use of 2-octylcyanoacrylate during repair of linear cutaneous surgery wounds improves scar cosmesis compared to wound closure with 5-0 fast absorbing gut.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the use of 2-octylcyanoacrylate during repair of linear cutaneous surgery wounds improves scar cosmesis compared to wound closure with 5-0 fast absorbing gut. The investigators will use a split wound model, where half of the wound is treated with 2-octylcyanoacrylate and the other half is repaired with 5-0 fast absorbing gut. Three-months post-surgery, the scar will be measured via the physician observer scar assessment scale, a validated scar instrument. The scar width, and adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure with predicted linear closure of 3 cm of longer.
* Willing to return for follow-up visits

Exclusion Criteria:

* Mentally handicapped
* Unable to understand written and oral English
* Incarceration
* Under 18 years of age
* Pregnant Women
* Wounds with predicted closure length less than 3 cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Assessment of Scar on the Patient and Observer Scar Assessment Scale | 3 months
  After surgical procedure, half of the subject's wound will be with 2-octylcyanoacrylate, while the other half is closed 5-0 fast absorbing gut sutures. After 3 months, subjects will return to clinic for evaluation of the cosmesis of both types of closure techniques.

SECONDARY OUTCOMES:
Measurement of Scar Width | 3 months
  The width of the scar will be measured 1 centimeter from the midline on both sides. There is no defined width that is considered satisfactory or not satisfactory. The measurements will be compared between subjects.
Assessment of Complications | 3 months
  Noting the presence or absence of bleeding, dehiscence, infection or spitting sutures.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, M.D., Principal Investigator — University of California, Davis

REFERENCES:
- [Derived] Zhuang AR, Beroukhim K, Armstrong AW, Sivamani RK, Eisen DB. Comparison of 2-Octylcyanoacrylate Versus 5-0 Fast-Absorbing Gut During Linear Wound Closures and the Effect on Wound Cosmesis. Dermatol Surg. 2020 May;46(5):628-634. doi: 10.1097/DSS.0000000000002076. PMID 31403536